CLINICAL TRIAL: NCT05205915
Title: Home-based Transcranial Direct Current Stimulation (tDCS) for Major Depressive Disorders (MDD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuroelectrics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NE02
Record Dates: First submitted 2021-12-20; First posted 2022-01-25 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm (Experimental): All patients will receive active treatment which consists of stimulation (tDCS) applied using the Starstim device, with current delivered via four Starstim Pi electrodes (circular electrodes with a contact of area of 3.14 cm2) embedded in the headpiece. All study subjects will use the same fixed montage (electrode locations and currents).
  Interventions: Device: tDCS intervention applied by Starstim device

INTERVENTIONS:
Device: tDCS intervention applied by Starstim device — Stimulation will be applied using the Starstim device, with current delivered via four Starstim Pi electrodes (circular electrodes with a contact of area of 3.14 cm2) embedded in the headpiece. All study subjects will use the same fixed montage (electrode locations and currents). The montage has been designed to optimize anodal stimulation in the desired target area while avoiding stimulation off target.
  Other Names: Starstim

SUMMARY:
This is an open label pilot feasibility telemedicine study. This pilot will involve a total of 37 at-home stimulation sessions (30-minutes each) of multichannel excitatory tDCS targeting the left dorsolateral prefrontal cortex (DLPFC) administered over 8 weeks, with a follow-up period of 4 weeks following the final stimulation session.

DETAILED DESCRIPTION:
This is an open label pilot feasibility telemedicine study. This pilot will involve a total of 37 at-home stimulation sessions (30-minutes each) of multichannel excitatory tDCS targeting the left dorsolateral prefrontal cortex (DLPFC) administered over 8 weeks, with a follow-up period of 4 weeks following the final stimulation session.

The main objective of the study is to assess the feasibility and safety of home-based tDCS for patients with MDD.

The treatment course will consist of an acute phase of 28 tDCS sessions, conducted daily (7 days per week) over 4 weeks.

Thereafter, participants will undergo a taper phase of an additional 9 sessions of tDCS applied in progressively decreasing frequency until day #60 of the study as follows:

1. Three tDCS sessions applied once every other day.
2. Three tDCS sessions applied once every third day.
3. Three tDCS sessions applied once every fourth day.

ELIGIBILITY:
Inclusion Criteria:

1. Major Depressive Disorder
2. Age >=18
3. Currently experiencing a major depressive episode of at least four weeks' duration
4. MADRS score at least 20 at trial entry.
5. Taking at least one approved antidepressant medication (except bupropion).
6. Has a healthcare provider, and a companion who can help administer study treatments; and be able to connect frequently with study staff
7. Access to wireless internet (wifi) connection

Exclusion Criteria:

1. Any psychotic disorder.
2. Concurrent benzodiazepine medication.
3. High suicide risk
4. History of significant neurological disorder.
5. Skin lesions on the scalp at the proposed electrode sites.
6. Pregnancy.
7. Any antidepressant medications will be permitted (except bupropion) provided the medication dose has been unchanged for 4 weeks prior to trial entry.
8. Any cranial metal implants (excluding ≤1 mm thick epicranial titanium skull plates and dental fillings) or
9. Medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagus nerve stimulator);
10. Previous surgeries opening the skull leaving skull defects capable of allowing the insertion of a cylinder with a radius greater or equal to 5 mm.
11. Substance use disorder (including alcohol) within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of incomplete and missed sessions (%) | From baseline to 4-week follow up across study subjects
  Feasibility will be evaluated using home-based data as recorded in the Neuroelectrics portal. Range [0,100]. Higher is worse
Incidence of Serious Adverse Events (SAE) | From baseline to 4-week follow up across study subjects
  Safety will be assessed by number and type of side effects
Median percentage change in Montgomery-Asberg Depression Mood Rating Scale (MADRS) scores | From baseline to 4-week follow up across study subjects
  The primary efficacy measure for this study will be the median percent change from baseline to the end of the 4-week post-treatment follow-up period in the observer-rated Montgomery-Asberg Depression Mood Rating Scale (MADRS) (Montgomery and Asberg, 1979). Range [0,100]. Higher is worse

SECONDARY OUTCOMES:
Response rate | From baseline to the 4-week follow-up
  Response rate is the secondary efficacy endpoint and will be calculated for the study subjects, where clinical response is defined as ≥ 50% improvement in Montgomery-Asberg Depression Mood Rating Scale (MADRS) score. Higher is better
Change in the Quick Inventory of Depressive Symptomatology (QIDS-SR) score | Change from baseline to 4-week follow-up in the participant-rated Quick Inventory of Depressive Symptomatology (QIDS-SR)
  Range [0,27]. Higher is worse
Change in the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) score | Change from baseline to 4-week follow-up in the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF)
  Range [14,70]. Higher is better
Median percentage change in Montgomery-Asberg Depression Mood Rating Scale (MADRS) scores | From baseline to the end of week 4 of treatment, and to the end of week 8 of treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Healthcare Innovations Institute, LLC, Coral Springs, Florida
  - Oceane7 Medical & Research Center, Inc., Miami, Florida
  - Renew Health Clinical Research, LLC, Snellville, Georgia
  - Conrad Clinical Research, Edmond, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ruffini G, Salvador R, Castaldo F, Baleeiro T, Camprodon JA, Chopra M, Cappon D, Pascual-Leone A. Multichannel tDCS with advanced targeting for major depressive disorder: a tele-supervised at-home pilot study. Front Psychiatry. 2024 Aug 15;15:1427365. doi: 10.3389/fpsyt.2024.1427365. eCollection 2024. PMID 39211540